CLINICAL TRIAL: NCT01872988
Title: Tenofovir Disoproxil Fumarate Improves Outcomes Following Palliative Transarterial Chemoembolization for Hepatitis B Virus Related Hepatocellular Carcinoma
Brief Title: Tenofovir Antiviral Therapy Following Transarterial Chemoembolization for HBV Related Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficult in patient enrollment
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Gilead Sciences (Industry); Taipei Institute of Pathology (Other Government)
Responsible Party: Principal Investigator, Chun-Ying Wu, Professor, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF12045; JIRB11-036-A (Other: JIRB, Taiwan)
Record Dates: First submitted 2013-01-30; First posted 2013-06-07 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Hepatitis B; Hepatocellular Carcinoma
Keywords: antiviral therapy; intermediate stage; hepatitis B virus
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular; Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir treatment (Active Comparator): Start to administer Tenofovir treatment 300mg PO QD within 2 weeks after the 1st TACE. Maximum duration of tenofovir treatment: 3 years.
  Interventions: Drug: Tenofovir
- Placebo (Placebo Comparator): Start to administer placebo 1 Tab PO QD within 2 weeks after the 1st TACE. Maximum duration of tenofovir treatment: 3 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenofovir — Administer Tenofovir to HCC patients who are indicated for TACE after randomization
  Other Names: Viread
  Arms: Tenofovir treatment
Drug: Placebo — Administer Placebo to HCC patients who are indicated for TACE after randomization
  Arms: Placebo

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common solid cancers worldwide, and chronic hepatitis B virus (HBV) infection is the most common etiology of HCC in Asia. Transarterial chemoembolization (TACE) is the standard treatment for patients with unresectable HCC in the BCLC intermediate stage, but the HCC recurrence rates and long-term mortality rates are quite high. These intermediate-staged HCC patients usually need repeated TACE due to tumor recurrence, and they may die of HCC progression or liver decompensation after repeated TACE. Improved liver function and decreased liver disease progression due to oral antiviral therapy have been proven to be effective for chronic hepatitis B, and oral antiviral therapy may keep better liver reserve and provide better chance for HCC patients received TACE. In addition, chronic HBV infection is one of the most important factors for HCC development, and antiviral therapy can improve the outcomes after curative treatment. However, the evidence of improving outcomes of HCC patients underwent TACE by oral antiviral therapy is lacking. Moreover, Tenofovir Disoproxil Fumarate (TDF) is one of the most potent oral antiviral agents, and its safety and very low long-term viral resistance rate have been also reported. There is no study to evaluate the impacts of TDF for HBV-related HCC patients underwent TACE. Until now, routine antiviral therapy for HBV-related HCC patients underwent TACE has still not been recommended by current guidelines. The hypothesis of this study is that a potent oral antiviral therapy for patients with HBV-related HCC patients receiving TACE improve patients' outcomes

DETAILED DESCRIPTION:
This is randomized double-blind placebo-controlled trial that will be conducted in referral teaching hospitals in Taiwan. This trial will recruit 320 patients fulfilling all of the following criteria: patients more than 20 years old, HCCs diagnosed by AASLD image criteria or pathology, medium-sized HCCs in BCLC intermediate stage and not more than 5 cm in maximum diameter and not more than 5 tumors that TACE is indicated, chronic HBV carrier (HBsAg+) with detectable HBV DNA in blood, ECOG performance status (PST) 0-2, Child-Pugh score ≦7, serum bilirubin < 2 mg/dL and prothrombin time (PT) prolongation < 3 seconds, and willingness to adhere to treatment and follow-up plans. Patients are ineligible if they have any of the following exclusion criteria: any vascular invasion by tumors, extra-hepatic metastasis, concurrent any other malignancy, concomitant immunosuppressive therapy, previous any HCC treatment, previous or current any antiviral therapy for HBV, concomitant other therapies for HCC except TACE, liver cirrhosis with severe gastroesophageal varices (EVF3 or with red color sign), poorly-controlled ascites or hepatic encephalopathy, contraindication for invasive procedures such as recent gastrointestinal bleeding or cerebral hemorrhage, contraindication to TACE such as allergy to contrast, pregnancy, sepsis, etc., chronic renal failure with eGFR < 60, concurrent any other chronic viral hepatitis with HCV, HDV, or HIV). The Primary endpoints of this study will be 1-, 3-year overall survival, and the secondary endpoints of this study will be time to tumor progression and time to liver decompensation.

ELIGIBILITY:
Inclusion Criteria:

1. more than 20 years old
2. HCCs diagnosed by AASLD image criteria or pathology
3. Intermediate-stage HCCs that TACE is indicated
4. chronic HBV carrier with detectable HBV DNA in blood
5. ECOG performance status (PST) 0-2
6. Child-Pugh score ≦7
7. serum bilirubin < 2 mg/dL
8. prothrombin time prolongation < 3 seconds
9. willingness to adhere to treatment and follow-up plans -

Exclusion Criteria:

1. any vascular invasion by tumors
2. extra-hepatic metastasis
3. concurrent any other malignancy
4. concomitant immunosuppressive therapy
5. HCC recurrence within 2 years of previous curative treatment
6. antiviral therapy for chronic hepatitis B within 6 months before HCC diagnosis
7. concomitant other therapies for HCC except TACE
8. liver cirrhosis with severe gastroesophageal varices (EVF3 or with red color sign), poorly-controlled ascites or hepatic encephalopathy
9. contraindication for invasive procedures such as recent gastrointestinal bleeding or cerebral hemorrhage
10. contraindication to TACE such as allergy to contrast, pregnancy, sepsis, etc.
11. chronic renal failure with eGFR < 60
12. concurrent any other chronic viral hepatitis with HCV, HDV, or HIV) -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 3-year

SECONDARY OUTCOMES:
time to tumor progression | 1- and 3-year
time to liver decompensation | 1- and 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ying Wu, MD, PhD, MPH, Principal Investigator — Taichung Veterans General Hospital; Jaw-Town Lin, MD, PhD, Study Chair — Fu Jen Catholic University
Locations (4):
- Taiwan (4):
  - Chia-Yi Christine Hospital, Chiayi City
  - E-Da Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Mackay Memorial Hosp, Taipei

REFERENCES:
- [Background] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766